CLINICAL TRIAL: NCT02140801
Title: A Randomised, Open-label, Parallel Group, Multi-center Study Using OCT to Comparing the Efficacy and Safety of Ticagrelor With Clopidogrel in the Prevention of Subclinical Thrombus in Patients After Drug-eluting Stent Implantation
Brief Title: Optical Coherence Tomography to Evaluate Ticagrelor and Clopidogrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISSBRIL0361
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Thrombosis
Keywords: Percutaneous coronary intervention; Drug-eluting stent; Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 90mg tablet, twice daily
  Interventions: Drug: Clopidogrel
- Clopidogrel (Experimental): Clopidogrel 75mg tablet, daily
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Plain, round, yellow, filmcoated tablet, 90 mg
  Other Names: BRILINTA™
  Arms: Clopidogrel
Drug: Clopidogrel — Orange brown capsule, containing one 75 mg clopidogrel tablet (cut into 2 halves)
  Other Names: Plavix®
  Arms: Ticagrelor

SUMMARY:
A number of 352 patients scheduled for elective percutaneous coronary intervention (PCI) with a native coronary stenosis suitable for DES implantation and OCT imaging are openly randomized 1:1 to either BRILINTA™ (ticagrelor) or Plavix® (clopidogrel bisulfate).

DETAILED DESCRIPTION:
The study is prospectively conducted at 4 high-volume PCI center in China with OCT expertise. Angiographic follow-up and OCT imaging with motorized pull-back at 20-36 mm/s are planned in all patients 12 months after implantation of the study stents. OCT endpoints are: (1) Subclinical intra-stent thrombus, defined as a mass protruding to the lumen with significant attenuation, and respectively (2) endothelial coverage, expressed as % of struts without coverage and % of stent length containing non-covered struts. The study is powered for OCT endpoints, which are likely to reach significance at the level P < 0.05 even at a follow-up drop-out rate up to 10%.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures;
* Men and women 18 years and older;.
* Established indication to PCI according to the guidelines of American Heart Association and American College of Cardiology;
* Native coronary lesion suitable for drug-eluting stent placement and OCT imaging.

Exclusion Criteria:

* Pregnancy and breast feeding mother;
* Co-morbidity with an estimated life expectancy of < 50 % at 12 months;
* Scheduled major surgery in the next 6 months;
* Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk;
* Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 30 days
* Cardiogenic shock
* Previous subacute or late coronary stent thrombosis
* Known allergy against ticagrelor, or against clopidogrel, or aspirin
* History of major hemorrhage (intracranial, gastrointestinal, etc.)
* Active pathological bleeding
* Acute or chronic hematologic disorder including a Hemoglobin less than 10 g/L or a platelet count less than 10×109/L before procedure
* Any history of Severe renal or hepatic dysfunction (hepatic failure, cirrhosis, portal hypertension and active hepatitis);
* Neutropenia,
* thrombocytopenia;
* Known acute pancreatitis
* Arterial aneurysm, arterial/venous malformation and aorta dissection.
* Culprit lesion within the proximal 10 mm of the right or left coronary artery
* Saphenous vein grafts
* Lesion length > 30 mm
* Involves a side branch ≥2.0 mm in diameter by visual estimate which requires treatment
* In-stent restenotic lesions
* Thombus-containing lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2014-05-01; Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Subclinical thrombus | 12 months
  The occurrence of subclinical thrombus as detected by OCT

SECONDARY OUTCOMES:
Endothelial coverage of the stent struts assessed by optical coherence tomography | 12 months
Neointimal proliferation within the stent assessed by optical coherence tomography | 12 months
Stent malposition assessed by optical coherence tomography | 12 months
Edge dissections assessed by optical coherence tomography | 12 months

OTHER OUTCOMES:
Bleeding events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Y, Wang YF, Zhao MY, You W, Xu T, Meng PN, Wu XQ, Wu ZM, Kong XH, Yin DL, Zhan ME, Jia HB, Liu B, Ye F. Study on the potential clinical significance of subclinical stent edge effects after drug-eluting stent implantation. Sci Rep. 2025 Mar 10;15(1):8258. doi: 10.1038/s41598-024-81329-7. PMID 40064903
- [Derived] Nong JC, You W, Wang YF, Xu Y, Xu T, Meng PN, Wu XQ, Wu ZM, Kong XH, Jia HB, Yin DL, Li L, Ye F. Dynamic natural components and morphological changes in nonculprit subclinical atherosclerosis in patients with acute coronary syndrome and mild chronic kidney disease at the 1-year follow-up and clinical significance at the 5-year follow-up. PLoS One. 2024 May 31;19(5):e0302547. doi: 10.1371/journal.pone.0302547. eCollection 2024. PMID 38820294
- [Derived] Meng PN, Nong JC, Xu Y, You W, Xu T, Wu XQ, Wu ZM, Tao BL, Guo YJ, Yin DL, Jia HB, Yang S, Ye F. Morphologies and composition changes in nonculprit subclinical atherosclerosis in diabetic versus nondiabetic patients with acute coronary syndrome who underwent long-term statin therapy. Sci Rep. 2023 Apr 1;13(1):5338. doi: 10.1038/s41598-023-32638-w. PMID 37005448
- [Derived] Nong JC, You W, Xu T, Meng PN, Xu Y, Wu XQ, Wu ZM, Tao BL, Guo YJ, Yang S, Yin DL, Ye F. Dynamic natural morphologies and component changes in nonculprit subclinical atherosclerosis in patients with acute coronary syndrome at 1-year follow-up and clinical significance at 3-year follow-up. Atherosclerosis. 2022 Sep;356:1-8. doi: 10.1016/j.atherosclerosis.2022.07.013. Epub 2022 Jul 31. PMID 35939981
- [Derived] Wu X, You W, Wu Z, Wu Q, Jiang J, Yan H, Ye F, Chen S. Ticagrelor versus clopidogrel for prevention of subclinical stent thrombosis detected by optical coherence tomography in patients with drug-eluting stent implantation-a multicenter and randomized study. Platelets. 2021 Apr 3;32(3):404-412. doi: 10.1080/09537104.2020.1754381. Epub 2020 Apr 24. PMID 32326796